CLINICAL TRIAL: NCT03224403
Title: A Randomized, Double-Blind, Placebo- and Active- Controlled, Single-Dose, Efficacy and Safety Study of a Test Acetaminophen 500 mg Tablet in Postoperative Dental Pain
Brief Title: Randomized, Double-Blind, Single-Dose, Efficacy and Safety Study of Test Acetaminophen Tablet in Postoperative Dental Pain
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Johnson & Johnson Consumer Inc., McNeil Consumer Healthcare Division (Industry)
Collaborators: Johnson & Johnson Consumer and Personal Products Worldwide (Industry)
Responsible Party: Sponsor
Organization: Johnson & Johnson Consumer and Personal Products Worldwide (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CO-170317095828-PACT
Record Dates: First submitted 2017-07-07; First posted 2017-07-21 (Actual); Results first posted 2021-04-15 (Actual); Last update posted 2021-04-15 (Actual); Status verified 2019-04

CONDITIONS: Post-operative Dental Pain

STUDY DESIGN:
Intervention Model Description: Post-operative dental pain following third molar extraction.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Test acetaminophen (Experimental): Test acetaminophen 1000 mg dose
  Interventions: Drug: Test acetaminophen
- Commercial acetaminophen (Active Comparator): Commercial acetaminophen 1000 mg dose
  Interventions: Drug: Commercial acetaminophen
- Commercial ibuprofen (Active Comparator): Commercial ibuprofen, 400 mg dose
  Interventions: Drug: Commercial ibuprofen
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Test acetaminophen — single dose of 2 Test acetaminophen 500 mg tablets
  Other Names: Test ACM
  Arms: Test acetaminophen
Drug: Commercial acetaminophen — single dose of 2 acetaminophen 500 mg caplets
  Other Names: Commercial ACM
  Arms: Commercial acetaminophen
Drug: Commercial ibuprofen — Single dose of 2 ibuprofen 200 mg Liquid-filled Capsules
  Other Names: Commercial IBU
  Arms: Commercial ibuprofen
Drug: Placebo — 2 placebo caplets
  Arms: Placebo

SUMMARY:
To evaluate analgesic onset, efficacy, and safety of 1000 mg acetaminophen administered as two Test Acetaminophen 500 mg tablets (Test ACM) compared with 1000 mg acetaminophen administered as two commercial acetaminophen 500 mg caplets (ACM) and 400 mg ibuprofen administered as two commercial ibuprofen 200 mg liquid-filled capsules (IBU) in the dental pain model following third-molar extractions.

DETAILED DESCRIPTION:
This is a single-dose, randomized, double-blind, placebo- and active- controlled, parallel-group study to evaluate the analgesic onset, efficacy, and safety profile of Test ACM 1000 mg compared with two commercial products over a four-hour period after third-molar extractions. Subjects will undergo dental extraction of three or four third molars.

ELIGIBILITY:
Inclusion Criteria:

1. 17 to 50 years old
2. Weigh 100 lbs. or greater and have a body mass index (BMI) of 18 to 30 (inclusive)
3. Dental extraction of three or four third molars
4. Meets post-surgical pain criteria
5. Females of childbearing age must be willing to use acceptable method of birth control

Exclusion Criteria:

1. Currently pregnant or planning to be pregnant or nursing a baby
2. Known allergy to acetaminophen, nonsteroidal anti-inflammatory drugs (NSAIDs) including aspirin, as well as hydrocodone or other opioids
3. Inability to swallow whole large tablets or capsules
4. Have other conditions that the investigator feels may impact subject's safety and/or the integrity of the study
5. Use of pain medications 5 or more times per week
6. Have a history of chronic tranquilizer use, heavy drinking, or substance abuse in the last 5 years
7. History of endoscopically documented peptic ulcer disease or bleeding disorder in the last 2 years
8. Have a positive urine drug screen

Ages: 17 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 664 (Actual)
Dates: Start 2017-07-19 (Actual); Primary Completion 2018-04-04 (Actual); Study Completion 2018-04-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Derek Muse, Principal Investigator — Jean Brown Research/ BB Holdings
Locations (1):
- Jean Brown Research, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: Yes
YODA

REFERENCES:
- [Derived] Myers A, Bertoch T, Zhang P, Cooper SA. Clinical validation of a fast-acting acetaminophen: a randomized, active and placebo controlled dental pain study. Curr Med Res Opin. 2024 May;40(5):839-848. doi: 10.1080/03007995.2024.2331159. Epub 2024 Mar 23. PMID 38505928
- [Derived] Myers A, Gelotte C, Zuckerman A, Zimmerman B, Shenoy A, Qi D, Cooper SA. Analgesic onset and efficacy of a fast-acting formulation of acetaminophen in a postoperative dental impaction pain model. Curr Med Res Opin. 2024 Feb;40(2):267-277. doi: 10.1080/03007995.2023.2294946. Epub 2024 Jan 24. PMID 38124555

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Two placebo caplets taken orally
- Test ACM 1000 mg: Two test acetaminophen 500 mg tablets taken orally
- Commercial ACM 1000 mg: Two commercial acetaminophen 500 mg caplets taken orally
- Commercial IBU 400 mg: Two commercial ibuprofen 200 mg liquid-filled capsules taken orally
Period: Overall Study
Arm/Group | Placebo | Test ACM 1000 mg | Commercial ACM 1000 mg | Commercial IBU 400 mg
Started | 59 | 249 | 232 | 124
Completed | 59 | 249 | 232 | 124
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Test ACM 1000 mg | Commercial ACM 1000 mg | Commercial IBU 400 mg | Total
Number analyzed (Participants) | 59 | 249 | 232 | 124 | 664
Age, Continuous [Mean (Standard Deviation); unit: years] | 18.3 (1.91) | 19.0 (2.31) | 18.9 (2.17) | 19.2 (2.56) | 18.9 (2.28)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 34 | 139 | 124 | 65 | 362
  Male | 25 | 110 | 108 | 59 | 302
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 1 | 1 | 1 | 4
  Asian | 0 | 3 | 3 | 5 | 11
  Native Hawaiian or Other Pacific Islander | 0 | 6 | 4 | 2 | 12
  Black or African American | 1 | 3 | 2 | 1 | 7
  White | 55 | 229 | 215 | 108 | 607
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 2 | 7 | 7 | 7 | 23
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 59 | 249 | 232 | 124 | 664

OUTCOME MEASURES:

1. Primary Outcome: Time to Confirmed Perceptible Pain Relief
Description: Minutes until confirmed perceptible pain relief is achieved. Stopwatch is started after the participant takes the study medication. The participant is instructed to stop the stopwatch when they first begin to feel any pain relief. The perceptible pain relief is confirmed if the participant also stopped the second stopwatch indicating meaningful pain relief.
Time Frame: within 4 hours
Population: Analysis is based on the Intent-to-Treat (ITT) population, which included all participants who were randomized.
Measure: Median (Full Range); unit: minutes
Arm/Group | Placebo | Test ACM 1000 mg | Commercial ACM 1000 mg | Commercial IBU 400 mg
Number analyzed (Participants) | 59 | 249 | 232 | 124
minutes | NA [4.9 to 240] — The median time to confirmed perceptible pain relief was not estimable since fewer than 50% of the participants treated with Placebo obtained confirmed perceptible pain relief. | 15.7 [2.2 to 240] | 20.2 [4 to 240] | 23.2 [2.5 to 240]
Statistical Analysis 1: Comparison: Placebo vs Test ACM 1000 mg; Test type: Superiority; p < 0.001, Wilcoxon test from SAS PROC LIFETEST — The significance threshold level was 0.049 (two-sided). P-values are based on the Wilcoxon test from PROC LIFETEST that compared survival curves
Statistical Analysis 2: Comparison: Placebo vs Commercial ACM 1000 mg; Test type: Superiority; p < 0.001, Wilcoxon test from SAS PROC LIFETEST — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Placebo vs Commercial IBU 400 mg; Test type: Superiority; p < 0.001, Wilcoxon test from SAS PROC LIFETEST — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 4: Comparison: Test ACM 1000 mg vs Commercial ACM 1000 mg; Test type: Superiority; p = 0.035, bootstrap re-sampling method — The significance threshold level was 0.049 (two-sided). P-values are from the comparison of median survival time using the bootstrap re-sampling method
Statistical Analysis 5: Comparison: Test ACM 1000 mg vs Commercial IBU 400 mg; Test type: Superiority; p < 0.001, bootstrap re-sampling method — [p-value comment as in outcome 1, analysis 4]

2. Secondary Outcome: Time to Meaningful Pain Relief
Description: Minutes until meaningful pain relief is achieved. Stopwatch is started after the participant takes the study medication. The participants are instructed to stop the stopwatch when the relief from the starting pain is meaningful to them.
Time Frame: Within 4 hours
Population: Analysis is based on the Intent-to-Treat (ITT) population, which included all participants who were randomized.
Measure: Median (Full Range); unit: minutes
Arm/Group | Placebo | Test ACM 1000 mg | Commercial ACM 1000 mg | Commercial IBU 400 mg
Number analyzed (Participants) | 59 | 249 | 232 | 124
minutes | NA [14.7 to 240] — The median time to meaningful pain relief was not estimable since fewer than 50% of the participants treated with this study medication obtained meaningful pain relief. | 46.1 [8.7 to 240] | 44.2 [12.6 to 240] | 43.9 [16.7 to 240]
Statistical Analysis 1: Comparison: Placebo vs Test ACM 1000 mg; Test type: Superiority; p < 0.001, Wilcoxon test from SAS PROC LIFETEST — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Placebo vs Commercial ACM 1000 mg; Test type: Superiority; p < 0.001, Wilcoxon test from SAS PROC LIFETEST — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Placebo vs Commercial IBU 400 mg; Test type: Superiority; p < 0.001, Wilcoxon test from SAS PROC LIFETEST — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 4: Comparison: Test ACM 1000 mg vs Commercial ACM 1000 mg; Test type: Superiority; p = 0.671, bootstrap re-sampling method — [p-value comment as in outcome 1, analysis 4]
Statistical Analysis 5: Comparison: Test ACM 1000 mg vs Commercial IBU 400 mg; Test type: Superiority; p = 0.487, bootstrap re-sampling method — [p-value comment as in outcome 1, analysis 4]

3. Secondary Outcome: Percentage of Participants With Confirmed Perceptible Relief From 30 Minutes to Successively Earlier Minutes in One-minute Increments - 30 Minutes
Description: Percentage of participants with confirmed perceptible relief by 30 minutes. Stopwatch is started after the participant takes the study medication. The participant is instructed to stop the stopwatch when they first begin to feel any pain relief. The perceptible pain relief is confirmed if the participant also stopped the second stopwatch indicating meaningful pain relief. Test acetaminophen 1000 mg and placebo were compared on the percentage of subjects with confirmed perceptible relief starting at 30 minutes and testing successively earlier minutes (29, 28, etc) until the difference was no longer statistically significant. The earliest significant time was identified.
Time Frame: by 30 minutes
Population: Analysis is based on the Intent-to-Treat (ITT) population, which included all participants who were randomized.
Measure: Number; unit: Percentage of Participants
Arm/Group | Placebo | Test ACM 1000 mg
Number analyzed (Participants) | 59 | 249
Percentage of Participants | 18.6 | 75.1
Statistical Analysis 1: Comparison: Placebo vs Test ACM 1000 mg; Test type: Superiority; p < 0.001, Regression, Logistic

4. Secondary Outcome: Percentage of Participants With Confirmed Perceptible Relief From 30 Minutes to Successively Earlier Minutes in One-minute Increments - 29 Minutes
Description: Percentage of participants with confirmed perceptible relief by 29 minutes. Stopwatch is started after the participant takes the study medication. The participant is instructed to stop the stopwatch when they first begin to feel any pain relief. The perceptible pain relief is confirmed if the participant also stopped the second stopwatch indicating meaningful pain relief. Test acetaminophen 1000 mg and placebo were compared on the percentage of subjects with confirmed perceptible relief starting at 30 minutes and testing successively earlier minutes (29, 28, etc) until the difference was no longer statistically significant. The earliest significant time was identified.
Time Frame: by 29 minutes
Population: Analysis is based on the Intent-to-Treat (ITT) population, which included all participants who were randomized.
Measure: Number; unit: Percentage of Participants
Arm/Group | Placebo | Test ACM 1000 mg
Number analyzed (Participants) | 59 | 249
Percentage of Participants | 18.6 | 73.5
Statistical Analysis 1: Comparison: Placebo vs Test ACM 1000 mg; Test type: Superiority; p < 0.001, Regression, Logistic

5. Secondary Outcome: Percentage of Participants With Confirmed Perceptible Relief From 30 Minutes to Successively Earlier Minutes in One-minute Increments - 28 Minutes
Description: Percentage of participants with confirmed perceptible relief by 28 minutes. Stopwatch is started after the participant takes the study medication. The participant is instructed to stop the stopwatch when they first begin to feel any pain relief. The perceptible pain relief is confirmed if the participant also stopped the second stopwatch indicating meaningful pain relief. Test acetaminophen 1000 mg and placebo were compared on the percentage of subjects with confirmed perceptible relief starting at 30 minutes and testing successively earlier minutes (29, 28, etc) until the difference was no longer statistically significant. The earliest significant time was identified.
Time Frame: by 28 minutes
Population: Analysis is based on the Intent-to-Treat (ITT) population, which included all participants who were randomized.
Measure: Number; unit: Percentage of Participants
Arm/Group | Placebo | Test ACM 1000 mg
Number analyzed (Participants) | 59 | 249
Percentage of Participants | 18.6 | 70.7
Statistical Analysis 1: Comparison: Placebo vs Test ACM 1000 mg; Test type: Superiority; p < 0.001, Regression, Logistic

6. Secondary Outcome: Percentage of Participants With Confirmed Perceptible Relief From 30 Minutes to Successively Earlier Minutes in One-minute Increments - 27 Minutes
Description: Percentage of participants with confirmed perceptible relief by 27 minutes. Stopwatch is started after the participant takes the study medication. The participant is instructed to stop the stopwatch when they first begin to feel any pain relief. The perceptible pain relief is confirmed if the participant also stopped the second stopwatch indicating meaningful pain relief. Test acetaminophen 1000 mg and placebo were compared on the percentage of subjects with confirmed perceptible relief starting at 30 minutes and testing successively earlier minutes (29, 28, etc) until the difference was no longer statistically significant. The earliest significant time was identified.
Time Frame: by 27 minutes
Population: Analysis is based on the Intent-to-Treat (ITT) population, which included all participants who were randomized.
Measure: Number; unit: Percentage of Participants
Arm/Group | Placebo | Test ACM 1000 mg
Number analyzed (Participants) | 59 | 249
Percentage of Participants | 18.6 | 70.7
Statistical Analysis 1: Comparison: Placebo vs Test ACM 1000 mg; Test type: Superiority; p < 0.001, Regression, Logistic

7. Secondary Outcome: Percentage of Participants With Confirmed Perceptible Relief From 30 Minutes to Successively Earlier Minutes in One-minute Increments - 26 Minutes
Description: Percentage of participants with confirmed perceptible relief by 26 minutes. Stopwatch is started after the participant takes the study medication. The participant is instructed to stop the stopwatch when they first begin to feel any pain relief. The perceptible pain relief is confirmed if the participant also stopped the second stopwatch indicating meaningful pain relief. Test acetaminophen 1000 mg and placebo were compared on the percentage of subjects with confirmed perceptible relief starting at 30 minutes and testing successively earlier minutes (29, 28, etc) until the difference was no longer statistically significant. The earliest significant time was identified.
Time Frame: by 26 minutes
Population: Analysis is based on the Intent-to-Treat (ITT) population, which included all participants who were randomized.
Measure: Number; unit: Percentage of Participants
Arm/Group | Placebo | Test ACM 1000 mg
Number analyzed (Participants) | 59 | 249
Percentage of Participants | 18.6 | 69.9
Statistical Analysis 1: Comparison: Placebo vs Test ACM 1000 mg; Test type: Superiority; p < 0.001, Regression, Logistic

8. Secondary Outcome: Percentage of Participants With Confirmed Perceptible Relief From 30 Minutes to Successively Earlier Minutes in One-minute Increments - 25 Minutes
Description: Percentage of participants with confirmed perceptible relief by 25 minutes. Stopwatch is started after the participant takes the study medication. The participant is instructed to stop the stopwatch when they first begin to feel any pain relief. The perceptible pain relief is confirmed if the participant also stopped the second stopwatch indicating meaningful pain relief. Test acetaminophen 1000 mg and placebo were compared on the percentage of subjects with confirmed perceptible relief starting at 30 minutes and testing successively earlier minutes (29, 28, etc) until the difference was no longer statistically significant. The earliest significant time was identified.
Time Frame: by 25 minutes
Population: Analysis is based on the Intent-to-Treat (ITT) population, which included all participants who were randomized.
Measure: Number; unit: Percentage of Participants
Arm/Group | Placebo | Test ACM 1000 mg
Number analyzed (Participants) | 59 | 249
Percentage of Participants | 18.6 | 69.5
Statistical Analysis 1: Comparison: Placebo vs Test ACM 1000 mg; Test type: Superiority; p < 0.001, Regression, Logistic

9. Secondary Outcome: Percentage of Participants With Confirmed Perceptible Relief From 30 Minutes to Successively Earlier Minutes in One-minute Increments - 24 Minutes
Description: Percentage of participants with confirmed perceptible relief by 24 minutes. Stopwatch is started after the participant takes the study medication. The participant is instructed to stop the stopwatch when they first begin to feel any pain relief. The perceptible pain relief is confirmed if the participant also stopped the second stopwatch indicating meaningful pain relief. Test acetaminophen 1000 mg and placebo were compared on the percentage of subjects with confirmed perceptible relief starting at 30 minutes and testing successively earlier minutes (29, 28, etc) until the difference was no longer statistically significant. The earliest significant time was identified.
Time Frame: by 24 minutes
Population: Analysis is based on the Intent-to-Treat (ITT) population, which included all participants who were randomized.
Measure: Number; unit: Percentage of Participants
Arm/Group | Placebo | Test ACM 1000 mg
Number analyzed (Participants) | 59 | 249
Percentage of Participants | 18.6 | 67.5
Statistical Analysis 1: Comparison: Placebo vs Test ACM 1000 mg; Test type: Superiority; p < 0.001, Regression, Logistic

10. Secondary Outcome: Percentage of Participants With Confirmed Perceptible Relief From 30 Minutes to Successively Earlier Minutes in One-minute Increments - 23 Minutes
Description: Percentage of participants with confirmed perceptible relief by 23 minutes. Stopwatch is started after the participant takes the study medication. The participant is instructed to stop the stopwatch when they first begin to feel any pain relief. The perceptible pain relief is confirmed if the participant also stopped the second stopwatch indicating meaningful pain relief. Test acetaminophen 1000 mg and placebo were compared on the percentage of subjects with confirmed perceptible relief starting at 30 minutes and testing successively earlier minutes (29, 28, etc) until the difference was no longer statistically significant. The earliest significant time was identified.
Time Frame: by 23 minutes
Population: Analysis is based on the Intent-to-Treat (ITT) population, which included all participants who were randomized.
Measure: Number; unit: Percentage of Participants
Arm/Group | Placebo | Test ACM 1000 mg
Number analyzed (Participants) | 59 | 249
Percentage of Participants | 18.6 | 66.3
Statistical Analysis 1: Comparison: Placebo vs Test ACM 1000 mg; Test type: Superiority; p < 0.001, Regression, Logistic

11. Secondary Outcome: Percentage of Participants With Confirmed Perceptible Relief From 30 Minutes to Successively Earlier Minutes in One-minute Increments - 22 Minutes
Description: Percentage of participants with confirmed perceptible relief by 22 minutes. Stopwatch is started after the participant takes the study medication. The participant is instructed to stop the stopwatch when they first begin to feel any pain relief. The perceptible pain relief is confirmed if the participant also stopped the second stopwatch indicating meaningful pain relief. Test acetaminophen 1000 mg and placebo were compared on the percentage of subjects with confirmed perceptible relief starting at 30 minutes and testing successively earlier minutes (29, 28, etc) until the difference was no longer statistically significant. The earliest significant time was identified.
Time Frame: by 22 minutes
Population: Analysis is based on the Intent-to-Treat (ITT) population, which included all participants who were randomized.
Measure: Number; unit: Percentage of Participants
Arm/Group | Placebo | Test ACM 1000 mg
Number analyzed (Participants) | 59 | 249
Percentage of Participants | 16.9 | 62.7
Statistical Analysis 1: Comparison: Placebo vs Test ACM 1000 mg; Test type: Superiority; p < 0.001, Regression, Logistic

12. Secondary Outcome: Percentage of Participants With Confirmed Perceptible Relief From 30 Minutes to Successively Earlier Minutes in One-minute Increments - 21 Minutes
Description: Percentage of participants with confirmed perceptible relief by 21 minutes. Stopwatch is started after the participant takes the study medication. The participant is instructed to stop the stopwatch when they first begin to feel any pain relief. The perceptible pain relief is confirmed if the participant also stopped the second stopwatch indicating meaningful pain relief. Test acetaminophen 1000 mg and placebo were compared on the percentage of subjects with confirmed perceptible relief starting at 30 minutes and testing successively earlier minutes (29, 28, etc) until the difference was no longer statistically significant. The earliest significant time was identified.
Time Frame: by 21 minutes
Population: Analysis is based on the Intent-to-Treat (ITT) population, which included all participants who were randomized.
Measure: Number; unit: Percentage of Participants
Arm/Group | Placebo | Test ACM 1000 mg
Number analyzed (Participants) | 59 | 249
Percentage of Participants | 15.3 | 60.2
Statistical Analysis 1: Comparison: Placebo vs Test ACM 1000 mg; Test type: Superiority; p < 0.001, Regression, Logistic

13. Secondary Outcome: Percentage of Participants With Confirmed Perceptible Relief From 30 Minutes to Successively Earlier Minutes in One-minute Increments - 20 Minutes
Description: Percentage of participants with confirmed perceptible relief by 20 minutes. Stopwatch is started after the participant takes the study medication. The participant is instructed to stop the stopwatch when they first begin to feel any pain relief. The perceptible pain relief is confirmed if the participant also stopped the second stopwatch indicating meaningful pain relief. Test acetaminophen 1000 mg and placebo were compared on the percentage of subjects with confirmed perceptible relief starting at 30 minutes and testing successively earlier minutes (29, 28, etc) until the difference was no longer statistically significant. The earliest significant time was identified.
Time Frame: by 20 minutes
Population: Analysis is based on the Intent-to-Treat (ITT) population, which included all participants who were randomized.
Measure: Number; unit: Percentage of Participants
Arm/Group | Placebo | Test ACM 1000 mg
Number analyzed (Participants) | 59 | 249
Percentage of Participants | 13.6 | 58.2
Statistical Analysis 1: Comparison: Placebo vs Test ACM 1000 mg; Test type: Superiority; p < 0.001, Regression, Logistic

14. Secondary Outcome: Percentage of Participants With Confirmed Perceptible Relief From 30 Minutes to Successively Earlier Minutes in One-minute Increments - 19 Minutes
Description: Percentage of participants with confirmed perceptible relief by 19 minutes. Stopwatch is started after the participant takes the study medication. The participant is instructed to stop the stopwatch when they first begin to feel any pain relief. The perceptible pain relief is confirmed if the participant also stopped the second stopwatch indicating meaningful pain relief. Test acetaminophen 1000 mg and placebo were compared on the percentage of subjects with confirmed perceptible relief starting at 30 minutes and testing successively earlier minutes (29, 28, etc) until the difference was no longer statistically significant. The earliest significant time was identified.
Time Frame: by 19 minutes
Population: Analysis is based on the Intent-to-Treat (ITT) population, which included all participants who were randomized.
Measure: Number; unit: Percentage of Participants
Arm/Group | Placebo | Test ACM 1000 mg
Number analyzed (Participants) | 59 | 249
Percentage of Participants | 13.6 | 56.2
Statistical Analysis 1: Comparison: Placebo vs Test ACM 1000 mg; Test type: Superiority; p < 0.001, Regression, Logistic

15. Secondary Outcome: Percentage of Participants With Confirmed Perceptible Relief From 30 Minutes to Successively Earlier Minutes in One-minute Increments - 18 Minutes
Description: Percentage of participants with confirmed perceptible relief by 18 minutes. Stopwatch is started after the participant takes the study medication. The participant is instructed to stop the stopwatch when they first begin to feel any pain relief. The perceptible pain relief is confirmed if the participant also stopped the second stopwatch indicating meaningful pain relief. Test acetaminophen 1000 mg and placebo were compared on the percentage of subjects with confirmed perceptible relief starting at 30 minutes and testing successively earlier minutes (29, 28, etc) until the difference was no longer statistically significant. The earliest significant time was identified.
Time Frame: by 18 minutes
Population: Analysis is based on the Intent-to-Treat (ITT) population, which included all participants who were randomized.
Measure: Number; unit: Percentage of Participants
Arm/Group | Placebo | Test ACM 1000 mg
Number analyzed (Participants) | 59 | 249
Percentage of Participants | 13.6 | 55.0
Statistical Analysis 1: Comparison: Placebo vs Test ACM 1000 mg; Test type: Superiority; p < 0.001, Regression, Logistic

16. Secondary Outcome: Percentage of Participants With Confirmed Perceptible Relief From 30 Minutes to Successively Earlier Minutes in One-minute Increments - 17 Minutes
Description: Percentage of participants with confirmed perceptible relief by 17 minutes. Stopwatch is started after the participant takes the study medication. The participant is instructed to stop the stopwatch when they first begin to feel any pain relief. The perceptible pain relief is confirmed if the participant also stopped the second stopwatch indicating meaningful pain relief. Test acetaminophen 1000 mg and placebo were compared on the percentage of subjects with confirmed perceptible relief starting at 30 minutes and testing successively earlier minutes (29, 28, etc) until the difference was no longer statistically significant. The earliest significant time was identified.
Time Frame: by 17 minutes
Population: Analysis is based on the Intent-to-Treat (ITT) population, which included all participants who were randomized.
Measure: Number; unit: Percentage of Participants
Arm/Group | Placebo | Test ACM 1000 mg
Number analyzed (Participants) | 59 | 249
Percentage of Participants | 13.6 | 53.8
Statistical Analysis 1: Comparison: Placebo vs Test ACM 1000 mg; Test type: Superiority; p < 0.001, Regression, Logistic

17. Secondary Outcome: Percentage of Participants With Confirmed Perceptible Relief From 30 Minutes to Successively Earlier Minutes in One-minute Increments - 16 Minutes
Description: Percentage of participants with confirmed perceptible relief by 16 minutes. Stopwatch is started after the participant takes the study medication. The participant is instructed to stop the stopwatch when they first begin to feel any pain relief. The perceptible pain relief is confirmed if the participant also stopped the second stopwatch indicating meaningful pain relief. Test acetaminophen 1000 mg and placebo were compared on the percentage of subjects with confirmed perceptible relief starting at 30 minutes and testing successively earlier minutes (29, 28, etc) until the difference was no longer statistically significant. The earliest significant time was identified.
Time Frame: by 16 minutes
Population: Analysis is based on the Intent-to-Treat (ITT) population, which included all participants who were randomized.
Measure: Number; unit: Percentage of Participants
Arm/Group | Placebo | Test ACM 1000 mg
Number analyzed (Participants) | 59 | 249
Percentage of Participants | 10.2 | 52.2
Statistical Analysis 1: Comparison: Placebo vs Test ACM 1000 mg; Test type: Superiority; p < 0.001, Regression, Logistic

18. Secondary Outcome: Percentage of Participants With Confirmed Perceptible Relief From 30 Minutes to Successively Earlier Minutes in One-minute Increments - 15 Minutes
Description: Percentage of participants with confirmed perceptible relief by 15 minutes. Stopwatch is started after the participant takes the study medication. The participant is instructed to stop the stopwatch when they first begin to feel any pain relief. The perceptible pain relief is confirmed if the participant also stopped the second stopwatch indicating meaningful pain relief. Test acetaminophen 1000 mg and placebo were compared on the percentage of subjects with confirmed perceptible relief starting at 30 minutes and testing successively earlier minutes (29, 28, etc) until the difference was no longer statistically significant. The earliest significant time was identified.
Time Frame: by 15 minutes
Population: Analysis is based on the Intent-to-Treat (ITT) population, which included all participants who were randomized.
Measure: Number; unit: Percentage of Participants
Arm/Group | Placebo | Test ACM 1000 mg
Number analyzed (Participants) | 59 | 249
Percentage of Participants | 10.2 | 41.4
Statistical Analysis 1: Comparison: Placebo vs Test ACM 1000 mg; Test type: Superiority; p < 0.001, Regression, Logistic

19. Secondary Outcome: Percentage of Participants With Confirmed Perceptible Relief From 30 Minutes to Successively Earlier Minutes in One-minute Increments - 14 Minutes
Description: Percentage of participants with confirmed perceptible relief by 14 minutes. Stopwatch is started after the participant takes the study medication. The participant is instructed to stop the stopwatch when they first begin to feel any pain relief. The perceptible pain relief is confirmed if the participant also stopped the second stopwatch indicating meaningful pain relief. Test acetaminophen 1000 mg and placebo were compared on the percentage of subjects with confirmed perceptible relief starting at 30 minutes and testing successively earlier minutes (29, 28, etc) until the difference was no longer statistically significant. The earliest significant time was identified.
Time Frame: by 14 minutes
Population: Analysis is based on the Intent-to-Treat (ITT) population, which included all participants who were randomized.
Measure: Number; unit: Percentage of Participants
Arm/Group | Placebo | Test ACM 1000 mg
Number analyzed (Participants) | 59 | 249
Percentage of Participants | 8.5 | 31.7
Statistical Analysis 1: Comparison: Placebo vs Test ACM 1000 mg; Test type: Superiority; p < 0.001, Regression, Logistic

20. Secondary Outcome: Percentage of Participants With Confirmed Perceptible Relief From 30 Minutes to Successively Earlier Minutes in One-minute Increments - 13 Minutes
Description: Percentage of participants with confirmed perceptible relief by 13 minutes. Stopwatch is started after the participant takes the study medication. The participant is instructed to stop the stopwatch when they first begin to feel any pain relief. The perceptible pain relief is confirmed if the participant also stopped the second stopwatch indicating meaningful pain relief. Test acetaminophen 1000 mg and placebo were compared on the percentage of subjects with confirmed perceptible relief starting at 30 minutes and testing successively earlier minutes (29, 28, etc) until the difference was no longer statistically significant. The earliest significant time was identified.
Time Frame: by 13 minutes
Population: Analysis is based on the Intent-to-Treat (ITT) population, which included all participants who were randomized.
Measure: Number; unit: Percentage of Participants
Arm/Group | Placebo | Test ACM 1000 mg
Number analyzed (Participants) | 59 | 249
Percentage of Participants | 8.5 | 25.7
Statistical Analysis 1: Comparison: Placebo vs Test ACM 1000 mg; Test type: Superiority; p = 0.007, Regression, Logistic

21. Secondary Outcome: Percentage of Participants With Confirmed Perceptible Relief From 30 Minutes to Successively Earlier Minutes in One-minute Increments - 12 Minutes
Description: Percentage of participants with confirmed perceptible relief by 12 minutes. Stopwatch is started after the participant takes the study medication. The participant is instructed to stop the stopwatch when they first begin to feel any pain relief. The perceptible pain relief is confirmed if the participant also stopped the second stopwatch indicating meaningful pain relief. Test acetaminophen 1000 mg and placebo were compared on the percentage of subjects with confirmed perceptible relief starting at 30 minutes and testing successively earlier minutes (29, 28, etc) until the difference was no longer statistically significant. The earliest significant time was identified.
Time Frame: by 12 minutes
Population: Analysis is based on the Intent-to-Treat (ITT) population, which included all participants who were randomized.
Measure: Number; unit: Percentage of Participants
Arm/Group | Placebo | Test ACM 1000 mg
Number analyzed (Participants) | 59 | 249
Percentage of Participants | 8.5 | 21.7
Statistical Analysis 1: Comparison: Placebo vs Test ACM 1000 mg; Test type: Superiority; p = 0.026, Regression, Logistic

22. Secondary Outcome: Percentage of Participants With Confirmed Perceptible Relief From 30 Minutes to Successively Earlier Minutes in One-minute Increments - 11 Minutes
Description: Percentage of participants with confirmed perceptible relief by 11 minutes. Stopwatch is started after the participant takes the study medication. The participant is instructed to stop the stopwatch when they first begin to feel any pain relief. The perceptible pain relief is confirmed if the participant also stopped the second stopwatch indicating meaningful pain relief. Test acetaminophen 1000 mg and placebo were compared on the percentage of subjects with confirmed perceptible relief starting at 30 minutes and testing successively earlier minutes (29, 28, etc) until the difference was no longer statistically significant. The earliest significant time was identified.
Time Frame: by 11 minutes
Population: Analysis is based on the Intent-to-Treat (ITT) population, which included all participants who were randomized.
Measure: Number; unit: Percentage of Participants
Arm/Group | Placebo | Test ACM 1000 mg
Number analyzed (Participants) | 59 | 249
Percentage of Participants | 8.5 | 18.1
Statistical Analysis 1: Comparison: Placebo vs Test ACM 1000 mg; Test type: Superiority; p = 0.080, Regression, Logistic

ADVERSE EVENTS:
Time Frame: Beginning with signing of the informed consent form and continuing within 7 days after dental surgery for non-serious adverse events, +30 days after the subject's last dose or exposure to the investigational product for serious adverse events.
Description: AEs were systematically collected during the study and at the follow-up telephone interview within 7 days after surgery along with spontaneously reported AEs. Any clinically important abnormalities or causally-related AEs persisting were followed until resolution or until reaching a clinically stable endpoint. SAEs required immediate notification to the Sponsor. Any SAE occurring after the reporting period was to be promptly reported if a causal relationship to study product was suspected.
Groups:
- Commercial ACM 1000 mg: Two test acetaminophen 500 mg tablets taken orally
- Commercial IBU 400 mg: Two commercial ibuprofen 400 mg liquid-filled capsules taken orally
Arm/Group | Placebo | Test ACM 1000 mg | Commercial ACM 1000 mg | Commercial IBU 400 mg
All-Cause Mortality (participants affected / at risk) | 0/59 | 0/249 | 0/232 | 0/124
Serious Adverse Events (participants affected / at risk) | 1/59 | 1/249 | 0/232 | 0/124
Other Adverse Events (participants affected / at risk) | 9/59 | 13/249 | 16/232 | 7/124
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=59) | Test ACM 1000 mg (N=249) | Commercial ACM 1000 mg (N=232) | Commercial IBU 400 mg (N=124)
Pyelonephritis (Infections and infestations) | 1 | 0 | 0 | 0
Abortion Spontaneous (Pregnancy, puerperium and perinatal conditions) | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=59) | Test ACM 1000 mg (N=249) | Commercial ACM 1000 mg (N=232) | Commercial IBU 400 mg (N=124)
Nausea (Gastrointestinal disorders) | 7 | 13 | 14 | 7
Vomiting (Gastrointestinal disorders) | 7 | 10 | 11 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol (2017-05-16): https://cdn.clinicaltrials.gov/large-docs/03/NCT03224403/Prot_000.pdf
  • Statistical Analysis Plan (2018-04-25): https://cdn.clinicaltrials.gov/large-docs/03/NCT03224403/SAP_001.pdf